CLINICAL TRIAL: NCT01163760
Title: Clinical Evaluation of Two Daily Disposable Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Collaborators: Singapore Polytechnic University (Unknown); Visioncare Research Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-0706; PRO-518
Record Dates: First submitted 2008-09-29; First posted 2010-07-16 (Estimated); Results first posted 2010-07-16 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2015-05

CONDITIONS: Refractive Error
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- etafilcon A / ocufilcon D (Other): etafilcon A contact lens worn first daily disposable , ocufilcon D contact lens worn second daily disposable
  Interventions: Device: etafilcon A; Device: ocufilcon D
- oculfilcon D / etafilcon A (Other): ocufilcon D contact lens worn first, etafilcon A contact lens worn second
  Interventions: Device: etafilcon A; Device: ocufilcon D
- ocufilcon D / ocufilcon D (Other): ocufilcon D contact lens worn first and second
  Interventions: Device: ocufilcon D
- etafilcon A / etafilcon A (Other): etafilcon A contact lens worn first and second
  Interventions: Device: etafilcon A

INTERVENTIONS:
Device: etafilcon A — daily disposable contact lens
  Arms: etafilcon A / etafilcon A; etafilcon A / ocufilcon D; oculfilcon D / etafilcon A
Device: ocufilcon D — daily disposable contact lens
  Arms: etafilcon A / ocufilcon D; ocufilcon D / ocufilcon D; oculfilcon D / etafilcon A

SUMMARY:
This study seeks to evaluate the clinical performance of two daily disposable contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Be between 21 and 39 years of age.
* Signed Written Informed Consent and Investigator to record this on Case Report Form (CRF) in appropriate space.
* Be existing (i.e. successfully worn for 1-month prior to the study) soft contact lens wearers (no extended wear in the last 3 months, but silicone hydrogels in daily wear are allowed).
* Require a visual correction in both eyes (monovision allowed but no monofit).
* Have a contact lens spherical distance requirement between -1.00D and -6.00D in both eyes.
* Astigmatism of 1.00D or less in both eyes.
* Be able to wear the lens powers available for this study.
* Be correctable to a visual acuity of 20/30 or better in each eye.
* Have normal eyes with no evidence of abnormality or disease. For the purposes of this study a normal eye is defined as one having:

  * No amblyopia.
  * No evidence of lid abnormality or infection.
  * No conjunctival abnormality or infection.
  * No clinically significant slit lamp findings (i.e. edema, staining, scarring, vascularisation, infiltrates or abnormal opacities).
  * No other active ocular disease.

Exclusion Criteria:

* Requires concurrent ocular medication.
* Any systemic illness which would contraindicate lens wear or the medical treatment of which would affect vision or successful lens wear.
* Clinically significant (Grade 3 or 4) corneal edema, corneal vascularisation, corneal staining, tarsal abnormalities, bulbar injection or any other abnormality of the cornea that would contraindicate contact lens wear.
* Diabetic.
* Infectious disease (e.g., hepatitis, tuberculosis) or an immunosuppressive disease (e.g., HIV).
* Extended lens wear in last 3 months.
* PMMA or RGP lens wear in the previous 8 weeks.
* Has had refractive surgery. Has had eye injury/surgery within 8 weeks immediately prior to enrollment for this study.
* Abnormal lacrimal secretions.
* Pre-existing ocular irritation that would preclude contact lens fitting.
* Keratoconus or other corneal irregularity.
* Pregnancy, lactating or planning a pregnancy at the time of enrollment.
* Participation in any concurrent clinical trial or in last 60 days."

Ages: 21 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2007-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 50 subjects enrolled in this single site study, located at Singapore University.
Pre-assignment Details: There were 50 patients enrolled and randomized, and 50 patients completed the study.
Groups:
- Etafilcon A First, Then Ocufilcon D: etafilcon A contact lenses worn first,ocufilcon D contact lenses worn second
- Ocufilcon D First, Then Etafilcon A: ocufilcon D contact lenses worn first,etafilcon A contact lenses worn second.
- Etafilcon A First, Then Etafilcon A: etafilcon A contact lenses worn for both periods.
- Ocufilcon D First, Then Ocufilcon D: Ocufilcon D contact lenses worn for both periods.
Period: Period 1 (Fit)
Arm/Group | Etafilcon A First, Then Ocufilcon D | Ocufilcon D First, Then Etafilcon A | Etafilcon A First, Then Etafilcon A | Ocufilcon D First, Then Ocufilcon D
Started | 12 | 13 | 13 | 12
Completed | 12 | 13 | 13 | 12
Not Completed | 0 | 0 | 0 | 0
Period: Period 2 (Follow-up)
Arm/Group | Etafilcon A First, Then Ocufilcon D | Ocufilcon D First, Then Etafilcon A | Etafilcon A First, Then Etafilcon A | Ocufilcon D First, Then Ocufilcon D
Started | 12 | 13 | 13 | 12
Completed | 12 | 13 | 13 | 12
Not Completed | 0 | 0 | 0 | 0
Period: Period 3 (Fit)
Arm/Group | Etafilcon A First, Then Ocufilcon D | Ocufilcon D First, Then Etafilcon A | Etafilcon A First, Then Etafilcon A | Ocufilcon D First, Then Ocufilcon D
Started | 12 | 13 | 13 | 12
Completed | 12 | 13 | 13 | 12
Not Completed | 0 | 0 | 0 | 0
Period: Period 4 (Follow-up)
Arm/Group | Etafilcon A First, Then Ocufilcon D | Ocufilcon D First, Then Etafilcon A | Etafilcon A First, Then Etafilcon A | Ocufilcon D First, Then Ocufilcon D
Started | 12 | 13 | 13 | 12
Completed | 12 | 13 | 13 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: Total number of completed participants are included in baseline measurements.
Arm/Group | Overall
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.0 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Lens Comfort
Description: Lens comfort was evaluated via the subjective question: "How comfortable did your eyes feel at the end of the day when wearing the contact lenses you were provided?" (excellent/very good=5...very good=3...Poor=0)
Time Frame: 1-week follow-up
Population: Subjects analyzed were those who were enrolled, randomized, and completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Etafilcon A: etafilcon A contact lenses worn in either the first or second period.
- Ocufilcon D: ocufilcon D contact lenses worn in either the first or second period.
Arm/Group | Etafilcon A | Ocufilcon D
Number analyzed (Participants) | 51 | 49
units on a scale | 3.08 (0.98) | 3.00 (1.15)

2. Secondary Outcome: Comfort Throughout the Whole Day
Description: Comfort throughout the day was evaluated via subjective question: "Comfort throughout the whole day" and is reported as an aggregate of "Agree Strongly and Agree Somewhat".
Time Frame: 1-week follow-up
Population: Subjects analyzed were those enrolled, randomized, and completed the study.
Measure: Number; unit: percentage of participants
Arm/Group | Etafilcon A | Ocufilcon D
Number analyzed (Participants) | 51 | 49
percentage of participants | 39.2 | 36.7

3. Other Pre Specified Outcome: Comfort While Working on Computer
Description: Comfort throughout the day was evaluated via subjective question: "Comfort while working on computer" and is reported as an aggregate of "Agree Strongly and Agree Somewhat".
Time Frame: 1-week-follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Etafilcon A | Ocufilcon D
Number analyzed (Participants) | 51 | 49
percentage of participants | 47.0 | 42.9

ADVERSE EVENTS:
Groups:
- Etafilcon A/ Ocufilcon D: etafilcon A contact lenses worn first,ocufilcon D contact lenses worn second
- Ocufilcon D / Etafilcon A: ocufilcon D contact lenses worn first,etafilcon A contact lenses worn second.
- Etafilcon A/ Etafilcon A: etafilcon A contact lenses worn first and second period.
- Oculfilcon D / Ocufilcon D: ocufilcon D contact lenses worn first and second period.
Arm/Group | Etafilcon A/ Ocufilcon D | Ocufilcon D / Etafilcon A | Etafilcon A/ Etafilcon A | Oculfilcon D / Ocufilcon D
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13 | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/13 | 0/13 | 0/12

LIMITATIONS AND CAVEATS:
The integrity of the subject reported data is suspect and not reflective of lens' performance due to a significant protocol deviation. Upon completion of the study it was found that subjects were unmasked and their data should be considered biased.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may not publish, divulge, reveal, disclose, or use the data and or results of the study without prior written consent of Vistakon.